CLINICAL TRIAL: NCT02947529
Title: The Use of Tranexamic Acid to Reduce the Need for Transfusion 1 Week Post-operatively for Hemiarthroplasty or Intramedullary Nailing Needed to Correct Acute Hip Fractures
Brief Title: Tranexamic Acid Use in Acute Hip Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Trevor Owen, MD, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD2016
Record Dates: First submitted 2016-10-13; First posted 2016-10-28 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Acute Hip Fractures
Keywords: Hemiarthroplasty; Intramedullary nail; Tranexamic acid; Transfusion
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects undergoing surgery for acute hip fractures with a long trochanteric femoral nail (TFN) or hemiarthroplasty will randomized 50:50 to receive 1 dose of either tranexamic acid (TXA) or saline placebo solution prior to surgery and 1 dose during wound closure.
Who Masked: Participant, Investigator
Masking Description: Both the participants and the operating surgeons, who are members of the investigative team, will be blinded to which study group the participant is in throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Hemiarthroplasty - Placebo (Placebo Comparator): Patients are placed into this arm based on the type of surgery performed and are randomized to receive placebo
  Interventions: Other: Placebo
- Intramedullary nail - Tranexamic Acid (Experimental): Patients are placed into this arm based on the type of surgery performed and are randomized to receive tranexamic acid
  Interventions: Drug: Tranexamic Acid
- Hemiarthroplasty - Tranexamic Acid (Experimental): Patients are placed into this arm based on the type of surgery performed and are randomized to receive tranexamic acid
  Interventions: Drug: Tranexamic Acid
- Intramedullary nail - Placebo (Placebo Comparator): Patients are placed into this arm based on the type of surgery performed and are randomized to receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — intravenous dose
  Other Names: TXA
  Arms: Hemiarthroplasty - Tranexamic Acid; Intramedullary nail - Tranexamic Acid
Other: Placebo — intravenous dose
  Other Names: Saline
  Arms: Hemiarthroplasty - Placebo; Intramedullary nail - Placebo

SUMMARY:
BACKGROUND: Tranexamic acid (TXA) has been used widely for the reduction of post operative blood loss for various orthopaedic procedures including but not limited to total hip arthroplasty and total knee arthroplasty. A recent multihospital meta-analysis conducted in 2013 showed that patients who received TXA showed a significant reduction in post-operative transfusion (20.1% to 7.7%). The procedures the investigators will be evaluating are the intramedullary nail for intertrochanteric fracture and hip hemiarthroplasty. These procedures are similar to the total hip or knee replacement in that they can result in significant blood loss that requires a post operative transfusion.

STUDY PURPOSE: To determine the efficacy of TXA to decrease the rate of post-operative transfusion for acute hip fractures repaired with the following two methods, intramedullary nailing for intertrochanteric fracture and hemiarthroplasty.

METHODS: The model for the study is a prospective randomized control trial. Patients will be placed in one of two arms of the study after passing our inclusion criteria. The arms will be for either the intramedullary nailing for intertrochanteric fracture or for hemiarthroplasty. These two categories will be subdivided into those receiving TXA and those not receiving TXA. The patients in each category will have standard post-operative care and laboratory testing. The investigators will record the patients in either arm of the study, whether it be no TXA or TXA, who require post-operative transfusion within 1 week of the operation.

DETAILED DESCRIPTION:
This is a prospective randomized control trial. Patients scheduled for either intramedullary nailing for intertrochanteric fractures or for hemiarthroplasty will be selected for the study population.

The proposed research is needed to bridge the gap between the efficacy of TXA in elective, non-emergency procedures (such as total knee arthoplasty and total hip arthroplasty) and its efficacy in emergent acute hip fracture interventions. This study will use intravenous TXA (1g pre-op and 1g post-op) to study its effect on both the reduction of blood loss during intramedullary nail for intertrochanteric fractures and hemiarthroplasty procedures, and the subsequent reduction in the rate of blood transfusion in this patient population.

Both study and control groups will have standard post-operative care and laboratory testing and will be followed for one year post-operatively to record adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients age 65 or older who require surgery for a low energy trauma hip fracture

Exclusion Criteria:

* Prothrombotic state
* Cardiac stent within the past year with corresponding antiplatelet therapy
* Mechanical heart valves
* Deep vein thrombosis history
* Aortic stenosis
* Currently on Coumadin
* Malignancy
* Kidney dialysis
* Non-English speaking patients
* Medications contraindicated with tranexamic acid.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Transfusion reduction rate | 1 week
  Determine the efficacy of Tranexamic Acid (TXA) in the reduction of allogenic blood transfusion within 1 week following either hemiarthroplasty or intramedullary nailing for intertrochanteric fracture.

SECONDARY OUTCOMES:
Tranexamic acid post operative complications | 1 year
  Determine what effect TXA has on post-operative complications within 1 year following surgery for either hemiarthroplasty or intramedullary nailing for intertrochanteric fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Owen, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poeran J, Rasul R, Suzuki S, Danninger T, Mazumdar M, Opperer M, Boettner F, Memtsoudis SG. Tranexamic acid use and postoperative outcomes in patients undergoing total hip or knee arthroplasty in the United States: retrospective analysis of effectiveness and safety. BMJ. 2014 Aug 12;349:g4829. doi: 10.1136/bmj.g4829. PMID 25116268